CLINICAL TRIAL: NCT04878393
Title: A Multi-centre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters and Safety Associated With the Use of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in Japan
Brief Title: A Research Study Looking at How Oral Semaglutide Works in People With Type 2 Diabetes in Japan, as Part of Local Clinical Practice
Acronym: PIONEER REAL
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4613; U1111-1247-5339 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Patients will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.

SUMMARY:
The purpose of the study is to collect information on how Rybelsus® works in people with type 2 diabetes and to see if Rybelsus® can lower their blood sugar levels, and to get side-effects information. Participants will get Rybelsus® as prescribed to them by the study doctor.

The study will last for about 8-10 months. Participants will be asked to complete a questionnaire about how they take their Rybelsus® tablets. Participants will complete this questionnaire during their normally scheduled visit with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Diagnosed with type 2 diabetes mellitus
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study
* Male or female, age above or equal to 20 years at the time of signing informed consent
* Available glycated haemoglobin (HbA1c) value greater than or equal to 90 days prior to the 'Informed Consent and Treatment Initiation visit' (Visit 1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (Visit 1) if in line with local clinical practice
* Treatment naïve to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than 14 days

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Treatment with any investigational drug within 30 days prior to enrolment into the study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  percent-points
Number of adverse event (AEs) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Count

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  percent
Absolute change in body weight | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Kilogram (Kg)
HbA1c less than 7 percent (Yes/No) | End of Study visit (Visit 3) (week 34-44)
  Percentage of patients achieving or not achieving the target value
HbA1c reduction greater than or equal to 1 percent-points and body weight reduction of greater than or equal to 5 percent (Yes/No) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Percentage of patients achieving or not achieving the target value
HbA1c reduction greater than or equal to 1 percent-points and body weight reduction of greater than or equal to 3 percent (Yes/No) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Percentage of patients achieving or not achieving the target value
Number of adverse reactions (ARs) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Count
Number of serious adverse events (SAEs) | From baseline (week 0) to End of Study visit (Visit3) (week 34-44)
  Count
Number of serious adverse reactions (SARs) | From baseline (week 0) to End of Study visit (Visit 3) (week 34-44)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Master Centre for Japan, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Suzuki R, Amadid H, Major-Pedersen A, Yabe D. PIONEER REAL Japan: Baseline characteristics of a multicenter, prospective, real-world study of oral semaglutide in adults with type 2 diabetes in clinical practice in Japan. J Diabetes Investig. 2024 Aug;15(8):1047-1056. doi: 10.1111/jdi.14219. Epub 2024 May 6. PMID 38711208